CLINICAL TRIAL: NCT05792085
Title: Heart Failure Optimization at Home to Improve Outcomes (Hozho): A Pragmatic Clinic Trial of Telephone-Based GDMT Optimization in Navajo Nation
Brief Title: Heart Failure Optimization at Home to Improve Outcomes (Hozho): A Pragmatic Clinical Trial in Navajo Nation
Acronym: Hozho
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Indian Health Service (IHS) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 02141989
Record Dates: First submitted 2023-01-26; First posted 2023-03-30 (Actual); Results first posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Stepped Wedge Design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth Model (Active Comparator): Patient enrolled in the GDMT Telehealth HF improvement program in which hone BP cuff is provided and medication is initiated and titrated over the phone
  Interventions: Behavioral: EHR-based GDMT Optimization
- Control (No Intervention): Usual care, control group

INTERVENTIONS:
Behavioral: EHR-based GDMT Optimization — Patients will be prescribed appropriate GDMT for HFrEF if they meet clinical criteria by the study team, appropriate lab work and follow up testing will be sent and followed up by the team. All recommendations and plans will be copied to primary care providers who can opt out if disagree, but also to improve telementoring to build clinical comfort.
  Arms: Telehealth Model

SUMMARY:
Heart failure causes significant morbidity and mortality, particularly in Navajo Nation. There are well-established evidence of improved mortality and lower heart failure hospitalizations with certain pharmacotherapies for heart failure with reduced ejection fraction (HFrEF). However, these medications are underutilized nationally, including in the Indian Health Service which is one important driver of poor heart failure outcomes. Therefore, as part of an EHR-based pragmatic clinic trial, we are implementing and testing a model that identifies American Indian HFrEF patients receiving care at one large Indian Health Service Site who meet clinical criteria for, but are not on appropriate therapy, and implements a model in patients are initiated and titrated on appropriate therapy over the phone with remote tele monitoring using home blood pressure cuff. We will evaluate the impact of this model to improve uptake of GDMT among HFrEF patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with heart failure with reduced ejection fraction with last ejection fraction equal to or less than 40%
* Have a primary care physician at Gallup Indian Medical Center or Tohatchi Health Center
* Have been seen in the last 12 months at Gallup Indian Medical Center or Tohatchi Health Center

Exclusion Criteria:

* On hospice
* LVAD/translant
* Home inotropes
* No visit in last 12 months at Gallup Indian Medical Center or Tohatchi Health Center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maricruz Merino, MD, Study Director — Indian Health Service (IHS); Lauren Eberly, MD, MPH, Principal Investigator — Indian Health Service, Upenn
Locations (2):
- United States (2):
  - Gallup Indian Medical Center, Gallup, New Mexico
  - Tohatchi Health Center, Tohatchi, New Mexico

IPD SHARING:
Plan to Share IPD: No
Patient data is protected by the Navajo Nation Human Research Board

REFERENCES:
- [Derived] Eberly LA, Tennison A, Mays D, Hsu CY, Yang CT, Benally E, Beyuka H, Feliciano B, Norman CJ, Brueckner MY, Bowannie C, Schwartz DR, Lindsey E, Friedman S, Ketner E, Detsoi-Smiley P, Shyr Y, Shin S, Merino M. Telephone-Based Guideline-Directed Medical Therapy Optimization in Navajo Nation: The Hozho Randomized Clinical Trial. JAMA Intern Med. 2024 Jun 1;184(6):681-690. doi: 10.1001/jamainternmed.2024.1523. PMID 38583185

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Patient enrolled in the GDMT Telehealth HF improvement program at t=0. in which home BP cuff is provided and medication is initiated and titrated over the phone with remote telemonitoring using a home BP cuff.
  Phone-based GDMT Optimization: Patients will be prescribed appropriate GDMT for HFrEF if they meet clinical criteria by the study team, appropriate lab work and follow up testing will be sent and followed up by the team. All recommendations and plans will be copied to primary care providers to build capacity and clinical comfort.
- Cohort 2: Remain in control group (usual care) from t=0 to t=30 days. At t=30 days, patients cross over into intervention arm and are enrolled in the GDMT Telehealth HF improvement program at t=30 days. in which home BP cuff is provided and medication is initiated and titrated over the phone with remote telemonitoring using a home BP cuff.
  Phone-based GDMT Optimization: Patients will be prescribed appropriate GDMT for HFrEF if they meet clinical criteria by the study team, appropriate lab work and follow up testing will be sent and followed up by the team. All recommendations and plans will be copied to primary care providers to build capacity and clinical comfort.
- Cohort 3: Remain in usual care from t=0 to t=60 days. At t=6- days, patients cross over into intervention arm and enrolled in the GDMT Telehealth HF improvement program at t=60 days. in which home BP cuff is provided and medication is initiated and titrated over the phone with remote telemonitoring using a home BP cuff.
  Phone-based GDMT Optimization: Patients will be prescribed appropriate GDMT for HFrEF if they meet clinical criteria by the study team, appropriate lab work and follow up testing will be sent and followed up by the team. All recommendations and plans will be copied to primary care providers to build capacity and clinical comfort.
- Cohort 4: Remain in usual care from t=0 to t=90 days. At t=90 days, patients cross over into intervention arm and enrolled in the GDMT Telehealth HF improvement program at t=90 days. in which home BP cuff is provided and medication is initiated and titrated over the phone with remote telemonitoring using a home BP cuff.
  Phone-based GDMT Optimization: Patients will be prescribed appropriate GDMT for HFrEF if they meet clinical criteria by the study team, appropriate lab work and follow up testing will be sent and followed up by the team. All recommendations and plans will be copied to primary care providers to build capacity and clinical comfort.
- Cohort 5: Remain in usual care from t=0 to t=120 days. At t=120 days, patients cross over into intervention arm and enrolled in the GDMT Telehealth HF improvement program at t=120 days. in which home BP cuff is provided and medication is initiated and titrated over the phone with remote telemonitoring using a home BP cuff.
  Phone-based GDMT Optimization: Patients will be prescribed appropriate GDMT for HFrEF if they meet clinical criteria by the study team, appropriate lab work and follow up testing will be sent and followed up by the team. All recommendations and plans will be copied to primary care providers to build capacity and clinical comfort.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Started | 21 | 21 (These patients eventually crossed over into the intervention in a stepped wedge design. Therefore, trial enrolled a total of 103 patients.) | 20 | 20 | 21
Completed | 21 | 21 | 20 | 20 | 20
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Arm/Group | Telehealth Model
Number analyzed (Participants) | 103
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65 [53 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 103
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 103
LVEF [Median (Inter-Quartile Range); unit: Percentage] | 32 [24 to 36]

OUTCOME MEASURES:

1. Primary Outcome: Percentage That Had Increase in Classes of Guideline Directed Medical Therapy
Description: % of Patients that had Increase in the number of classes of Guideline Directed Medical Therapy (Beta-blocker, ACEi/Angiotensin receptor blockers, Angiotensin Receptor-Neprilysin Inhibitor, Aldosterone receptor antagonists, SGLT2i)
Time Frame: 30 days
Measure: Number; unit: percentage of patients
Arm/Group | Telehealth Model | Control
Number analyzed (Participants) | 102 | 82
percentage of patients | 66.2 | 13.1

2. Secondary Outcome: Percentage That Had Increase in Classes of Guideline Directed Medical Therapy or Dose of Guideline Directed Medical Therapy
Description: Proportion of patients that had an increase in the number of classes or dose of Guideline Directed Medical Therapy (Beta-blocker, Angiotensin-converting enzyme inhibitors/Angiotensin receptor blockers, Angiotensin Receptor-Neprilysin Inhibitor, Aldosterone receptor antagonists, Sodium-glucose co-transporter 2 inhibitors)
Time Frame: 30 days
Measure: Number; unit: percentage of patients
Arm/Group | Telehealth Model | Control
Number analyzed (Participants) | 102 | 81
percentage of patients | 79 | 22.6

3. Secondary Outcome: Rates of Increase/Addition of ACEi/ARB/Angiotensin Receptor-Neprilysin Inhibitor
Description: Rates of Rx for ACEi, ARB, or ANRI (Sacubritril-Valsartan)
Time Frame: 30 days
Measure: Number; unit: Percentage of patients
Groups:
- Telehealth Model: Patient enrolled in the GDMT Telehealth HF improvement program in which home BP cuff is provided and medication is initiated and titrated over the phone
  EHR-based GDMT Optimization: Patients will be prescribed appropriate GDMT for HFrEF if they meet clinical criteria by the study team, appropriate lab work and follow up testing will be sent and followed up by the team. All recommendations and plans will be copied to primary care providers who can opt out if disagree, but also to improve telementoring to build clinical comfort.
Arm/Group | Telehealth Model | Control
Number analyzed (Participants) | 102 | 81
Percentage of patients | 39.7 | 6.3

4. Secondary Outcome: Rates of Increase/Addition in Sodium-glucose Co-transporter 2 Inhibitors
Description: Rates of Rx for Sodium-glucose co-transporter 2 inhibitors
Time Frame: 30 days
Measure: Number; unit: Percentage of patients
Arm/Group | Telehealth Model | Control
Number analyzed (Participants) | 102 | 81
Percentage of patients | 37.2 | 4.6

5. Secondary Outcome: Rates of Increase/Addition of Aldosterone Receptor Antagonists
Description: Rates of Rx for Aldosterone receptor antagonists
Time Frame: 30 days
Measure: Number; unit: Percentage of patients
Arm/Group | Telehealth Model | Control
Number analyzed (Participants) | 102 | 81
Percentage of patients | 30.6 | 0.9

6. Secondary Outcome: Rates of Increase/Addition of Beta-blockers
Description: Rates of Rx for Beta-blockers
Time Frame: 30 days
Measure: Number; unit: Percentage of patients
Arm/Group | Telehealth Model | Control
Number analyzed (Participants) | 102 | 81
Percentage of patients | 3.5 | 2.1

7. Secondary Outcome: Addition of or Increase in Dose for ACEi/ARB/ARNI
Description: Increase in Dose for ACEi/ARB/ARNI
Time Frame: 30 days
Measure: Number; unit: Percentage of patients
Arm/Group | Telehealth Model | Control
Number analyzed (Participants) | 102 | 81
Percentage of patients | 46.7 | 8.8

8. Secondary Outcome: Addition of or Increase in Dose of Beta-blocker
Description: Addition of or Increase in Dose for Beta-blocker
Time Frame: 30 days
Measure: Number; unit: Percentage of patients
Arm/Group | Telehealth Model | Control
Number analyzed (Participants) | 102 | 81
Percentage of patients | 17.4 | 8

9. Secondary Outcome: Addition of or Increase in Dose of Aldosterone Receptor Antagonists
Description: Dose increase or addition of Aldosterone receptor antagonists
Time Frame: 30 days
Measure: Number; unit: Percentage of patients
Arm/Group | Telehealth Model | Control
Number analyzed (Participants) | 102 | 81
Percentage of patients | 38.4 | 6.5

10. Other Pre Specified Outcome: Change in Provider Comfort With Guideline Directed Medical Therapy Prescribing From Baseline to 6 Months
Description: Baseline and follow up comfort prescribing therapy: Through survey we will assess at baseline and on follow-up how comfortable (from 1-5) providers feel with prescribing each of the following medications: Beta-blocker, Aldosterone receptor antagonist, Angiotensin-converting enzyme inhibitors, Angiotensin Receptor-Neprilysin Inhibitors, Sodium-glucose co-transporter 2 inhibitors. This measure is a score on a scale from 1-5, with 1 indicating low comfort level and 5 indicating high comfort level.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline: Provider survey of comfort pre-implementation of the model (at baseline)
- 6 Months: Provider comfort post-implementation of telehealth model (6 months)
Arm/Group | Baseline | 6 Months
Number analyzed (Participants) | 27 | 27
score on a scale | 1.86 (0.86) | 4.36 (0.63)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Cohort 1: Patients in cohort 1 receive the intervention (telehealth model) immediately (t=0 days) while the other cohorts (1-4) remain in usual care.
- Cohort 2: Patients in cohort 2 are randomized to receive the intervention at t=30 days. Patients in cohort 2 receive usual care until t=30 days when they cross over to receive the intervention (telehealth model) (t=30 days) while the other cohorts (3-5) remain in usual care.
- Cohort 3: Patients in cohort 3 are randomized to receive the intervention at t=60 days. Patients in cohort 3 receive usual care until t=60 days when they cross over to receive the intervention (telehealth model) (t=60 days) while the other cohorts (4-5) remain in usual care.
- Cohort 4: Patients in cohort 4 are randomized to receive the intervention at t=90 days. Patients in cohort 4 receive usual care until t=90 days when they cross over to receive the intervention (telehealth model) (t=90 days) while cohort 5 remains in usual care.
- Cohort 5: Patients in cohort 5 are randomized to receive the intervention at t=120 days. Patients in cohort 5 receive usual care until t=120 days when they cross over to receive the intervention (telehealth model) (t=120days).
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21 | 0/20 | 1/20 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/20 | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 2/21 | 3/21 | 2/20 | 4/20 | 8/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=21) | Cohort 2 (N=21) | Cohort 3 (N=20) | Cohort 4 (N=20) | Cohort 5 (N=21)
Any other minor adverse event (Cardiac disorders) | 2 (2) | 3 | 2 | 4 | 8 — Minor adverse events including hyperkalemia, hypokalemia, hyponatremia, acute kidney injury (creatinine increase >0.3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-06): https://cdn.clinicaltrials.gov/large-docs/85/NCT05792085/Prot_SAP_000.pdf